CLINICAL TRIAL: NCT00344474
Title: A New School-based Drug Prevention Programme for Teenagers: Interventions That Target Personality Risk for Substance Abuse and Mental Illness
Brief Title: Personality-targeted Interventions for Adolescent Alcohol Misuse
Acronym: Preventure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Action on Addiction (Other)
Responsible Party: Patricia J. Conrod, King's College London
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: PAJTXVA; 229/03
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2006-02

CONDITIONS: Alcohol Abuse; Drug Abuse; Depression; Panic Disorder; Conduct Disorder
Keywords: Prevention; Addiction; Personality; Adolescents; Binge Drinking; Alcohol Abuse; Comorbidity; Depression; Anxiety; Antisocial Behaviour
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Depression; Panic Disorder; Conduct Disorder; Behavior, Addictive; Binge Drinking; Anxiety Disorders; Antisocial Personality Disorder

ARMS (4):
- learning to cope with your impulsivity (Experimental): cognitive behavioural intervention teaching high impulsive youth how to manage their impulsive thinking and behaviours
  Interventions: Behavioral: PRE-Venture: Personality Risk Education
- learning to cope with your sensation seeking (Experimental): cognitive-behavioural intervention teaching high sensation seeking youth how to manage their need for stimulation and excitement
  Interventions: Behavioral: PRE-Venture: Personality Risk Education
- learning to cope with your anxiety sensitivity (Experimental): cognitive behavioural intervention targeting catastrophic thinking in high anxiety sensitive youth
  Interventions: Behavioral: PRE-Venture: Personality Risk Education
- learning to manage your negative thinking (Experimental): cognitive behavioural intervention targeting pessimistic and negative thinking in hopeless youth
  Interventions: Behavioral: PRE-Venture: Personality Risk Education

INTERVENTIONS:
Behavioral: PRE-Venture: Personality Risk Education — Motivational and Cognitive-Behavioural interventions targeting four personality risk factors for substance misuse. Two, 90-minute group sessions conducted at school with personality-matched peers and trained psychologists/councellors and co-facilitators.

SUMMARY:
Personality targeted cognitive behavioural interventions have been shown to be effective in reducing alcohol and drug misuse in adult substance abusers (Conrod et al., 2000) and adolescent drinkers (Conrod et al, in press). As these interventions target personality traits linked to risk for addictive and non-addictive mental disorders, the aim of this study is to examine the extent to which this approach can prevent and/or reduce alcohol and drug misuse as well as have an impact on the onset or severity of emotional and behavioural problems in young people.

DETAILED DESCRIPTION:
Personality targeted cognitive behavioural interventions have been shown to be effective in reducing alcohol and drug misuse in adult substance abusers (Conrod et al., 2000) and adolescent drinkers (Conrod et al, in press). As these interventions target personality traits linked to risk for addictive and non-addictive psychopathology, the aim of this study is to examine the extent to which this approach is effective in preventing and/or reduce alcohol and drug misuse and concurrent psychiatric symptoms in young people.

Method: 875 Participants aged 13-16 years will be screened for personality risk in school-wide self-report assessments. Participants will be randomly assigned to a personality matched cognitive-behavioural intervention or a no-intervention control. The personality matched interventions will target four personality risk factors: negative thinking (NT), anxiety sensitivity (AS), impulsivity (IMP) and sensation seeking (SS). Outcome evaluation will occur 6, 12, 18 and 24 months post intervention. Primary outcomes will be time to onset and severity of alcohol and illicit substance use and misuse. Secondary outcome variables will include depressive symptoms, panic attack rates, reckless and antisocial behaviour. Secondary analyses involving genetic, cognitive and coping skills measures will examine moderators of treatment effects.

Hypotheses: It is expected that personality-targeted interventions will have personality-specific effects on aspects of addictive and non-addictive psychopathology to which each personality risk group is most susceptible.

ELIGIBILITY:
Inclusion Criteria:

* secondary school student
* scoring one standard deviation above the school mean on one of 4 personality dimensions.
* Able to provide consent from parent/guardian for participation in the study

Exclusion Criteria:

* None

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 710 (Actual)
Dates: Start 2003-11; Primary Completion 2006-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Time to onset and severity of drug use | 2 years
  time to illicit drug use events, assessed using the Reckless Behaviour Questionnaire
Frequency and Quantity of Drinking | 2 years
Problem drinking symptoms | 2 years
  Assessed using an abbreviated version of the Rutger's Alcohol Problem Index

SECONDARY OUTCOMES:
Psychiatric symptoms (depression, panic anxiety, antisocial behaviours), coping skills, motives for drinking | 2 years
  Assessed using the Brief Symptom Inventory, the Reckless Behaviour Questionnaire, and the Drinking Motives Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J. Conrod, Ph.D., Principal Investigator — Institute of Psychiatry
Locations (1):
- Institute of Psychiatry, King's College London, London, United Kingdom

REFERENCES:
- [Background] Stewart SH, Conrod PJ, Marlatt GA, Comeau MN, Thush C, Krank M. New developments in prevention and early intervention for alcohol abuse in youths. Alcohol Clin Exp Res. 2005 Feb;29(2):278-86. doi: 10.1097/01.alc.0000153547.34399.e8. PMID 15714051
- [Background] Conrod PJ, Pihl RO, Stewart SH, Dongier M. Validation of a system of classifying female substance abusers on the basis of personality and motivational risk factors for substance abuse. Psychol Addict Behav. 2000 Sep;14(3):243-56. doi: 10.1037//0893-164x.14.3.243. PMID 10998950
- [Background] Conrod PJ, Stewart SH, Pihl RO, Cote S, Fontaine V, Dongier M. Efficacy of brief coping skills interventions that match different personality profiles of female substance abusers. Psychol Addict Behav. 2000 Sep;14(3):231-42. doi: 10.1037//0893-164x.14.3.231. PMID 10998949
- [Background] Comeau N, Stewart SH, Loba P. The relations of trait anxiety, anxiety sensitivity, and sensation seeking to adolescents' motivations for alcohol, cigarette, and marijuana use. Addict Behav. 2001 Nov-Dec;26(6):803-25. doi: 10.1016/s0306-4603(01)00238-6. PMID 11768546
- [Derived] Edalati H, Afzali MH, Castellanos-Ryan N, Conrod PJ. The Effect of Contextual Risk Factors on the Effectiveness of Brief Personality-Targeted Interventions for Adolescent Alcohol Use and Misuse: A Cluster-Randomized Trial. Alcohol Clin Exp Res. 2019 May;43(5):997-1006. doi: 10.1111/acer.14016. Epub 2019 Apr 8. PMID 30865304
- [Derived] Topper LR, Castellanos-Ryan N, Mackie C, Conrod PJ. Adolescent bullying victimisation and alcohol-related problem behaviour mediated by coping drinking motives over a 12 month period. Addict Behav. 2011 Jan-Feb;36(1-2):6-13. doi: 10.1016/j.addbeh.2010.08.016. Epub 2010 Sep 24. PMID 20869813
- [Derived] O'Leary-Barrett M, Mackie CJ, Castellanos-Ryan N, Al-Khudhairy N, Conrod PJ. Personality-targeted interventions delay uptake of drinking and decrease risk of alcohol-related problems when delivered by teachers. J Am Acad Child Adolesc Psychiatry. 2010 Sep;49(9):954-963.e1. doi: 10.1016/j.jaac.2010.04.011. Epub 2010 Jul 31. PMID 20732631
- [Derived] Conrod PJ, Castellanos-Ryan N, Strang J. Brief, personality-targeted coping skills interventions and survival as a non-drug user over a 2-year period during adolescence. Arch Gen Psychiatry. 2010 Jan;67(1):85-93. doi: 10.1001/archgenpsychiatry.2009.173. PMID 20048226